CLINICAL TRIAL: NCT03776071
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 3 Study of Enzastaurin Added to Temozolomide During and Following Radiation Therapy in Newly Diagnosed Glioblastoma Patients Who Possess the Novel Genomic Biomarker DGM1
Brief Title: A Trial of Enzastaurin Plus Temozolomide During and Following Radiation Therapy in Patients With Newly Diagnosed Glioblastoma With or Without the Novel Genomic Biomarker, DGM1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Denovo Biopharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DB102-01
Record Dates: First submitted 2018-12-12; First posted 2018-12-14 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RT plus TMZ and ENZ; ENZ alone; TMZ and ENZ (Active Comparator): Radiotherapy (RT) plus temozolomide (TMZ) and enzastaurin (ENZ) (Concurrent Phase) followed by enzastaurin alone (Single-Agent Phase), then temozolomide and enzastaurin (Adjuvant Phase)
  Interventions: Drug: Enzastaurin Hydrochloride; Drug: Temozolomide; Radiation: Radiotherapy
- RT plus TMZ and placebo; placebo; TMZ and placebo (Placebo Comparator): Radiotherapy (RT) plus temozolomide (TMZ) and placebo followed placebo then by temozolomide and placebo
  Interventions: Other: Placebo; Drug: Temozolomide; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Enzastaurin Hydrochloride — mg
  Other Names: Kinenza
  Arms: RT plus TMZ and ENZ; ENZ alone; TMZ and ENZ
Other: Placebo — mg
  Arms: RT plus TMZ and placebo; placebo; TMZ and placebo
Drug: Temozolomide — mg/m^2
  Other Names: Temodar
Radiation: Radiotherapy — Gy

SUMMARY:
This study will be conducted as a randomized, double-blind, placebo-controlled, multi-center Phase 3 study. Approximately 300 subjects with newly diagnosed glioblastoma who meet all eligibility criteria will be enrolled.

ELIGIBILITY:
Patient Inclusion Criteria:

Patients must meet all the following inclusion criteria to be eligible for enrollment into the study:

1. Signed informed consent
2. Age ≥ 18 years with life expectancy > 12 weeks
3. Histologically proven, newly diagnosed supratentorial glioblastoma (IDH mutant is excluded) based on the WHO classification (2016) which includes gliosarcoma (GS); prior diagnosis of lower grade astrocytoma that has been upgraded to histologically confirmed glioblastoma is eligible if chemotherapy and radiation therapy treatment-naïve
4. Randomization must occur within approximately 6 weeks after resection (patients undergoing biopsy only are excluded from the study)
5. Craniotomy site must be adequately healed, free of drainage or cellulitis and the underlying cranioplasty must appear intact prior to start of study treatment
6. DGM1 biomarker status (positive or negative) is available prior to randomization
7. Availability of tumor tissue representative of glioblastoma from surgery, and MGMT promoter methylation status is determined prior to study randomization
8. Karnofsky performance status (KPS) ≥ 70 (Appendix 1)
9. Stable or decreasing corticosteroids within 5 days prior to study treatment start
10. Willing to forego the use of Tumor Treating Fields therapy (Optune®)
11. Adequate organ function within 14 days prior to randomization:

    Bone marrow
    1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L;
    2. Platelet count ≥ 100 x 109/L;
    3. Hemoglobin ≥ 10 g/dL (eligibility level for hemoglobin may be met by transfusion) Renal
    4. Serum creatinine < 1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min as calculated using an appropriately validated prediction equation for the estimation of eGFR (eg, Cockcroft-Gault or MDRD method).

       Hepatic
    5. Total serum bilirubin ≤ 1.5 x ULN unless the patient has documented Gilbert syndrome;
    6. Aspartate and Alanine transaminase (AST/SGOT and ALT/SGPT) ≤ 2.5 x ULN;
    7. Alkaline phosphatase (ALP) ≤ 2.5 x ULN
12. Negative serum pregnancy test (for females of childbearing potential) within 7 days prior to the first study treatment
13. Male and female patients of reproductive potential must agree to use an effective method of contraception (eg, oral contraceptives, intrauterine device, barrier method) throughout the study and for at least 3 months after the last dose of study treatment, or 6 months for female patients in regard to the last dose of temozolomide (TMZ), whichever is later

    * Men are considered of reproductive potential unless they have undergone a vasectomy and confirmed sterile by a post-vasectomy semen analysis
    * Male patients must agree not to donate their semen during treatment with temozolomide and for at least 6 months after their last dose of temozolomide
    * Women are considered of reproductive potential unless they have undergone hysterectomy and/or surgical sterilization (at least 6 weeks following a bilateral oophorectomy, bilateral tubal ligation, or bilateral tubal occlusive procedure that has been confirmed in accordance with the device's label), have medically confirmed ovarian failure, or achieved postmenopausal status (defined as cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by having a serum follicle-stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal women
14. Willing and able to comply with the protocol

Patient Exclusion Criteria:

Patients with any of the following characteristics/conditions will be excluded from study:

1. Unable to swallow tablets or capsules
2. Pregnant or breastfeeding
3. Prior chemotherapy (including carmustine-containing wafers (Gliadel®), immunotherapy (including vaccine therapy), or investigational products for GBM or GS (previous 5-aminolevulinic acid (ALA)-mediated photodynamic therapy (PDT) administered prior to surgery to aid in optimal surgical resection is permitted)
4. Glioblastoma IDH mutant
5. Prior radiation therapy to the brain
6. Unable to discontinue use of enzyme-inducing anti-epileptic drugs (EIAEDs), see Section 5.1.2.4.1; if previously taking EIAEDs, must have been discontinued ≥ 2 weeks prior to randomization
7. Use of a strong inducer or moderate or strong inhibitor of CYP3A4 (Appendix 2) within 7 days prior to randomization or expected requirement for use on study therapy
8. Use of warfarin that cannot be stopped prior to the study.
9. Use of any medication that can prolong the QT/QTc interval (Appendix 3) within 7 days prior to start of study therapy, or plan to use such a medication during the study
10. Active bacterial, fungal or viral infection requiring systemic treatment
11. Personal or family history of abnormal long QT interval, QTc interval > 450 msec (males) or > 470 msec (females) as read on the printout of the electrocardiogram (ECG) at screening (recommended that QTc be calculated using Fridericia's correction formula, QTcF: see Section 7.3.2.2), or a history of unexplained syncope
12. Unstable angina; myocardial infarction or coronary artery bypass graft/percutaneous stent placement within 6 months of starting study treatment, congestive heart failure requiring treatment (New York Heart Association [NYHA] Grade ≥2)
13. History of significant cardiac arrhythmia (ventricular tachycardia or fibrillation, Torsades de Pointe) or second- or third-degree A-V block, symptomatic bradycardia (unless controlled with a pacemaker)
14. Persistent electrolyte abnormalities such as hypokalemia or hypomagnesemia that do not respond to treatment
15. History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)
16. Evidence of chronic hepatitis C infection as indicated by antibody to hepatitis C virus (HCV) with positive HCV ribonucleic acid (RNA)
17. Evidence of active or chronic hepatitis B infection as indicated by either:

    hepatitis B surface antigen (HBsAg) positive, or hepatitis B core antibody (HBcAb) positive with hepatitis B virus-deoxyribonucleic acid (HBV-DNA) positive (any detectable amount is considered positive)
18. Any contraindication to temozolomide listed in the local product label
19. Another malignancy except adequately treated non-melanoma skin cancer; patients who have had another primary malignancy in the past, but have been disease-free for more than 5 years, and patients who have had a localized malignancy treated with curative intent and disease free for more than 2 years are eligible
20. Participation in other studies involving investigational product(s) within 30 days prior to randomization
21. Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Up to 3 years

CONTACTS AND LOCATIONS:
Locations (65):
- United States (47):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic - Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center - Duarte, Duarte, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Irvine Health Chao Family Comprehensive Cancer Center, Orange, California
  - The University of Southern California, Pasadena, California
  - University of California San Francisco Helen Diller Family Comprehensive CA Ctr, San Francisco, California
  - University of Colorado Hospital Anschutz Cancer Pavilion, Aurora, Colorado
  - Blue Sky Neurology, Englewood, Colorado
  - Smilow Cancer Hospital - New Haven, New Haven, Connecticut
  - Lynn Cancer Institute, Boca Raton, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kentucky Markey Cancer Center, Lexington, Kentucky
  - Norton Cancer Institute - Multidisciplinary Clinic, Louisville, Kentucky
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - John Nasseff Neuroscience Institute, Minneapolis, Minnesota
  - Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine Center for Advanced Medicine, St Louis, Missouri
  - Hackensack Meridian Health - JFK Medical Center, Edison, New Jersey
  - New York University Medical Oncology Associates, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - New York - Presbyterian - Weill Cornell Medical Center, New York, New York
  - Messino Cancer Centers, Asheville, North Carolina
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health - Comprehensive Cancer Center, Winston-Salem, North Carolina
  - The Ohio State University - The James Cancer Hospital and Solove Research Institute, Columbus, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Penn Medicine - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - SCRI - Tennessee Oncology - Nashville - Centennial, Nashville, Tennessee
  - Vanderbilt - Ingram Cancer Center, Nashville, Tennessee
  - Austin Cancer Center - Park St. David's, Austin, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Lynn Cancer Institute, Houston, Texas
  - University of Texas Health Science Center at Houston (UT Health), Houston, Texas
  - Mays Cancer Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Canada (6):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Abbotsford, Abbotsford, British Columbia
  - British Columbia Cancer Agency - Victoria, Victoria, British Columbia
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Hôpital Fleurimont, Sherbrooke, Quebec
  - Saskatoon Cancer Center, Saskatoon, Saskatchewan
- China (12):
  - First Affiliated Hospital of USTC - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Tian Tan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Sanbo Brain Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Tongji Hospital, Wuhan, Hubei
  - Shengjing Hospital - Nanhu Campus, Shenyang, Liaoning
  - Tangdu Hospital, Xi'an, Shaanxi
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - General Hospital of Tianjin Medical University, Tianjin, Tianjin Municipality
  - Tianjin Huanhu Hospital, Xianshuigu, Tianjin Municipality